CLINICAL TRIAL: NCT04972266
Title: European Hypotension Prediction Index Real World Experience Using AcumenTM Hypotension Prediction Index Software to Prevent Intraoperative Hypotension: the Multicentre Prospective Observational Registry
Brief Title: The EU Hyprotect Registry
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Collaborators: IPPMed - Institut für Pharmakologie und Präventive Medizin GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-08
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-01

CONDITIONS: Hemodynamic Monitoring
Keywords: Intraoperative hypotension, Preventive Therapy, Blood pressure monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: AcumenTM Hypotension Prediction Index software — The AcumenTM HPI Feature Software provides the clinician with physiological insight into a patient's likelihood of trending toward a hypotensive event. The AcumenTM HPI Feature Software suite is enabled by the minimally invasive Acumen IQ sensor.

SUMMARY:
European, multicenter, prospective, observational registry in patients undergoing elective major non-cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients (≥18 years)
* Patient is scheduled for elective major non-cardiac surgery under general anesthesia that is expected to last at least 120 minutes and in whom blood pressure is monitored using an arterial catheter
* Patients in whom the AcumenTM Hypotension Prediction Index software with the Acumen IQ sensor on the Hemosphere platform is used intraoperatively

Exclusion Criteria:

* Patients undergoing emergency surgery OR nephrectomy, liver and/or kidney transplantation
* Patients suffering from atrial fibrillation and/or sepsis (according to current Sepsis-3 definition)
* American Society of Anesthesiology (ASA) physical status classification V or VI
* Disability and/or other circumstances under which the patient is not able to understand the nature, significance and scope of the investigation
* Pregnancy at the time of surgery
* Patients without signed informed consent / data protection statement
* Patient participating in other interventional trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elective major non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
To describe the time-weighted average (TWA) mean arterial pressure (MAP) <65 mmHg when using AcumenTM Hypotension Prediction Index software | Duration of the procedure through 30 days after procedure
  To describe the time-weighted average (TWA) mean arterial pressure (MAP) <65 mmHg when using AcumenTM Hypotension Prediction Index software

CONTACTS AND LOCATIONS:
Locations (12):
- France (2):
  - Hôpital Lariboisière, Paris
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (4):
  - Marien Hospital Herne, University Hospital Ruhr-University Bochum, Herne, Rhine-Westphalia
  - Justus Liebig University Giessen, University Hospital of Giessen and Marburg, Giessen
  - University Medical Center Hamburg Eppendorf, Hamburg
  - University Hospital Philipps-Universität Marburg, University Hospital of Giessen and Marburg, Marburg
- Italy (3):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti "Umberto I° General, Ancona
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona, Ancona
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Spain (2):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
- York and Scarborough Teaching Hospitals NHS Foundation Trust, Clifton, York, United Kingdom

IPD SHARING:
Plan to Share IPD: No